CLINICAL TRIAL: NCT01509664
Title: Encouraging Healthy Food Shopping and Eating Behaviors by Price Reduction: A Community Supermarket Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Obesity and Nutrition Research Center (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Dr. Allan Geliebter, Principal Investigator, New York Obesity and Nutrition Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-115
Record Dates: First submitted 2012-01-03; First posted 2012-01-13 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Discount intervention (Experimental): Receives 50% discount intervention on selected fruits and vegetables at participating supermarket.
  Interventions: Behavioral: Discount intervention
- Control (No Intervention): Received no discount at the participating supermarket.

INTERVENTIONS:
Behavioral: Discount intervention — 50% discount on selected fruits and vegetables at participating supermarket
  Arms: Discount intervention

SUMMARY:
The investigators plan to test the effect of price reduction of fruits and vegetables and non-caloric beverages on food purchasing, food intake, body weight, and body composition of primarily single adult shoppers. One hundred subjects will be randomized to an experimental or control group for a 4 month period. In the experimental group, there will be an automated 50% reduction in fruits vegetables and non-caloric beverages during the middle 2-month period. The investigators expect to observe significant changes in food shopping and eating behavior during this period, which should lead to body weight and fat loss. Some of these new shopping patterns should persist in the last month of the study even though prices revert.

ELIGIBILITY:
Inclusion Criteria:

* regularly buy 50% of groceries at designated supermarket
* primary food shopper for household, shopping for up to one other person, not counting children ≤ 6 years old

Exclusion Criteria:

* significant medical or psychiatric conditions
* participation in a weight loss program or a related study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2006-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — New York Obesity and Nutrition Research Center
Locations (1):
- St. Luke's Roosevelt Hospital center, New York, New York, United States

REFERENCES:
- [Background] Bernales-Korins M, Ang IYH, Khan S, Geliebter A. Psychosocial Influences on Fruit and Vegetable Intake Following a NYC Supermarket Discount. Obesity (Silver Spring). 2017 Aug;25(8):1321-1328. doi: 10.1002/oby.21876. Epub 2017 Jun 7. PMID 28590084
- [Result] Geliebter A, Ang IYH, Bernales-Korins M, Hernandez D, Ochner CN, Ungredda T, Miller R, Kolbe L. Supermarket discounts of low-energy density foods: effects on purchasing, food intake, and body weight. Obesity (Silver Spring). 2013 Dec;21(12):E542-8. doi: 10.1002/oby.20484. Epub 2013 Jul 5. PMID 23596089
- See also: New York Obesity and Nutrition Research Center — http://www.nyorc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via advertisement
Period: Overall Study
Arm/Group | Discount Intervention | Control
Started | 49 | 49
T2 Follow-up | 45 | 38
T3 Follow-up | 40 | 33
Completed | 34 | 28
Not Completed | 15 | 21
Not completed — Lost to Follow-up | 15 | 21

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Discount Intervention | Control | Total
Number analyzed (Participants) | 34 | 28 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (14) | 41 (14) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 7 | 32
  Male | 9 | 21 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 26 | 19 | 45
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 30 | 25 | 55
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Gross Weekly Purchasing of Fruits and Vegetables
Description: Gross weekly purchasing of fruits and vegetables from the discounted items list in $
Time Frame: week
Measure: Mean (Standard Error); unit: $
Arm/Group | Discount Intervention | Control
Number analyzed (Participants) | 34 | 28
$ | 5.57 (3.26) | 1.79 (2.06)

ADVERSE EVENTS:
Time Frame: Adverse Event Reporting data were collected whilst participants were actively participating in study procedures
Arm/Group | Discount Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/28
Other Adverse Events (participants affected / at risk) | 0/34 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No